CLINICAL TRIAL: NCT00725595
Title: Treatment of Cheyne Stocks Respiration With Adaptive Servo Ventilation and Bilevel Ventilators in Patients With Chronic Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Glenn Richard, ResMed Inc. of Australia
Other Study IDs: 092801; 20070928; No 092801
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2008-08-26 (Estimated); Status verified 2008-08

CONDITIONS: Heart Failure; Sleep Apnea
Keywords: Cheyne Stocks respiration; heart failure; sleep apnea; ventilator
MeSH Terms: conditions — Heart Failure; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- E, 2, III: To treat CSR with ASV and Bilevel ventilators

SUMMARY:
The overall purpose of this study is to determine the effects of adaptive servo ventilation (ASV) and bi-level ventilators on Cheyne-Stocks respiration (CSR). CSR is a pattern of breathing characterized by hyperpneas followed by hypopneas and or apneas. Clinically, the physiologic changes translate to sleep fragmentation, excessive daytime sleepiness, reduced exercise capacity and possibly ventricular arrhythmias. The intent of the proposed intervention is to compare the efficacies of ASV and Bi-level ventilator on CSR.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or legal representative of the patient is willing and able to sign an IRB/MEC approved informed consent and Privacy Protection Authorization in the United States
2. Subject is > 18 years old
3. Patients with known history of CSR. CSR symptoms may include the following:

   * sleep fragmentation as reported by patient or as witnessed by another person
   * night arousal after apneic episodes
   * reduced exercise capacity
   * daytime sleepiness
4. Expected to tolerate the ventilator therapy

Exclusion Criteria:

1. Baseline oxygen saturation < 90% on a stable FIO2)
2. Patient is currently enrolled in another clinical study which may confound the results of this study
3. Patient for whom informed consent cannot be obtained
4. Patient who is of pregnant or of child bearing potential without a negative pregnancy test within 10 days of the study procedure
5. Patients implanted with unable to tolerate inactive pacemaker, implantable defibrillator or cardiac resynchronization device for duration of testing procedure - approximately 8 hours (e.g. pacemaker dependency)
6. Patients with severe COPD (per GOLD scale)
7. Patients with a history of myocardial infarction within the 6 months prior to the study
8. Patients with unstable angina

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with both CSR and heart failure
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2008-08; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Both ASV and Bilevel ventilation are effective in clinical treatment of CSR | three months

SECONDARY OUTCOMES:
ASV treatment is more effective in removal or reduction of Cheyne-Stocks respiration than Bilevel ventilator for patients with chronic heart failure | three months

CONTACTS AND LOCATIONS:
Locations (1):
- The 1st Affiliated Hospitak of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Result] Zhang XL, Yin KS, Jiang SS, Li XL, Jia EZ, Su M. [Efficacy of adaptive pressure support servo-ventilation in patients with congestive heart failure and Cheyne-Stokes respiration]. Zhonghua Yi Xue Za Zhi. 2006 Jun 20;86(23):1620-3. Chinese. PMID 16854301